CLINICAL TRIAL: NCT01270841
Title: A Randomized, Double Blind, Placebo and Active Controlled, Parallel, Multi-Center Phase IIb Study to Evaluate Normalization of Morning Testosterone Levels in Men With Secondary Hypogonadism
Brief Title: Normalization of Morning Testosterone Levels in Men With Secondary Hypogonadism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZA-203
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-06

CONDITIONS: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; Enclomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Testim (topical testosterone) (Active Comparator): Testim (topical testosterone)
  Interventions: Drug: topical testosterone
- Androxal 12.5 mg (Experimental): Androxal 12.5 mg/day
  Interventions: Drug: Androxal
- Androxal 25 mg (Experimental): Androxal 25 mg/day
  Interventions: Drug: Androxal

INTERVENTIONS:
Drug: Placebo — Placebo capsule 1x daily for 3 months
  Arms: Placebo
Drug: topical testosterone — testosterone gel applied 1x daily for 3 months
  Other Names: Testim; AndroGel
  Arms: Testim (topical testosterone)
Drug: Androxal — Capsule of either 12.5 mg or 25 mg Androxal, 1x daily for 3 months
  Other Names: Enclomiphene citrate
  Arms: Androxal 12.5 mg; Androxal 25 mg

SUMMARY:
The Purpose of the study is to determine the effects of Androxal on morning testosterone and reproductive status in men with secondary hypogonadism(confirmed morning Testosterone less than 250 ng/dL), compared to changes with placebo, or Testim (topical testosterone). The effects of Testim versus placebo on reproductive status will also be examined. Study subjects must not be currently using a topical testosterone.

DETAILED DESCRIPTION:
This study is a phase IIb, 4 arm study with three month active dosing period. Three of the four treatment groups will be randomized to either Androxal or placebo in a double-blind fashion, and the fourth treatment group will receive open-label Testim. The doses of Androxal in the blinded portion of the study will be 12.5 mg and 25 mg, in capsule form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males between the ages of 21 and 65 years of age
* All clinical laboratory tests within normal ranges (any clinically significant deviation of laboratory results will require approval of sponsor)
* Previously or concurrently diagnosed as having secondary hypogonadism and confirmed morning testosterone <250ng/dL (two assessments at least 10 days apart)
* Ability to complete the study in compliance with the protocol
* Ability to understand and provide written informed consent
* Agreement to use double barrier contraception if with a fertile female partner
* Agreement to provide a semen sample in the clinic

Exclusion Criteria:

* Use of an injectable, oral, topical, or subcutaneous pelleted testosterone within 6 months prior to study
* Use of spironolactone, cimetidine, Clomid, 5α-reductase inhibitors, hCG, androgen, estrogen, anabolic steroid, DHEA, or herbal hormone products during the study
* Use of Clomid in the past year
* Uncontrolled hypertension or diabetes mellitus based on the Investigator's assessment at baseline. Subjects treated for Type II diabetes but exhibiting glycemic control will be allowed into the study
* A hematocrit >50% or a hemoglobin >17 g/dL
* Clinically significant abnormal findings on screening examination
* Use of an investigational drug or product, or participation in a drug or medical device research study within 30 days prior to receiving study medication
* Known hypersensitivity to Clomid
* Symptomatic cataracts (nuclear sclerosis cataract or cortical cataract grade > 2 based on 0-4 scale or any trace of posterior subcapsular cataract)
* Any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he took part in the study
* Irreversibly infertile or compromised fertility (cryptorchism, Kallman Syndrome, primary hypogonadism, vasectomy, or tumors of the pituitary)
* Current or history of breast cancer
* Current or history of prostate cancer or a suspicion of prostate disease unless ruled out by prostate biopsy, or a PSA>3.6
* Presence or history of hyperprolactinemia with or without a tumor
* Chronic use of medications use such as glucocorticoids
* Subjects with cystic fibrosis (mutation of the CFTR gene)
* Subjects unable to provide a semen sample in the clinic
* Subject has a BMI >36 kg/m2

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Lipshultz, MD, Principal Investigator — Baylor College of Medicine
Locations (18):
- United States (18):
  - Paradigm Clinical Inc., Garden Grove, California
  - Northern California Research Corp, Sacramento, California
  - Medical Center for Clinical Research, San Diego, California
  - Los Angeles Biomedical Research Institute, Torrance, California
  - Affiliated Clinical Research, Las Vegas, Nevada
  - Affiliated Clinical Research Inc., Las Vegas, Nevada
  - Weill Cornell Medical College and Smith Institute, Great Neck, New York
  - Jed Kaminetsky, New York, New York
  - Natan Bar-Chama, New York, New York
  - Michael A Werner, Purchase, New York
  - Discovery Clinical Trials, Austin, Texas
  - Research Across America, Carrollton, Texas
  - Texas Urology Specialist, Houston, Texas
  - Centex Research, Houston, Texas
  - Endocrine and Psychiatry Center, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - R/D Clinical Research, Lake Jackson, Texas
  - Cetero Research, San Antonio, Texas

REFERENCES:
- [Derived] Wiehle RD, Fontenot GK, Wike J, Hsu K, Nydell J, Lipshultz L; ZA-203 Clinical Study Group. Enclomiphene citrate stimulates testosterone production while preventing oligospermia: a randomized phase II clinical trial comparing topical testosterone. Fertil Steril. 2014 Sep;102(3):720-7. doi: 10.1016/j.fertnstert.2014.06.004. Epub 2014 Jul 17. PMID 25044085
- See also: Sponsor website — http://www.reprosrx.com
- See also: Website — http://www.helpmylowT.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Testim (Topical Testosterone) | Androxal 12.5 mg | Androxal 25 mg
Started | 29 | 33 | 29 | 33
Completed | 16 | 19 | 18 | 20
Not Completed | 13 | 14 | 11 | 13
Not completed — Adverse Event | 0 | 1 | 0 | 3
Not completed — Withdrawal by Subject | 3 | 2 | 3 | 3
Not completed — Lost to Follow-up | 3 | 1 | 4 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Did not qualify | 6 | 3 | 4 | 5
Not completed — Protocol Violation | 1 | 5 | 0 | 0
Not completed — Enrolled in error | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Testim (Topical Testosterone) | Androxal 12.5 mg | Androxal 25 mg | Total
Number analyzed (Participants) | 28 | 33 | 27 | 33 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (11.7) | 52.0 (10.6) | 49.7 (11.6) | 49.2 (10.9) | 50.6 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 28 | 33 | 27 | 33 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1 | 2
  Asian | 4 | 6 | 2 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 7 | 4 | 5 | 6 | 22
  White | 17 | 23 | 18 | 20 | 78
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 33 | 27 | 33 | 121
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.9 (4.2) | 33.1 (5.9) | 32.6 (5.2) | 31.7 (4.9) | 32.1 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Morning Testosterone
Description: Changes in values from baseline in total morning testosterone levels at month 3 comparing Androxal 12.5 and 25 mg to placebo and Testim
Time Frame: 3 months
Population: Intent to treat subjects with an assessment after baseline
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Placebo | Testim (Topical Testosterone) | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 26 | 30 | 25 | 32
ng/dL | -16.9 (47.5) | 253.7 (292.3) | 258.5 (201.5) | 197.3 (162.6)

2. Secondary Outcome: Change in Luteinizing Hormone Levels
Description: Changes in values from baseline in LH at month 3
Time Frame: 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Placebo | Testim (Topical Testosterone) | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 26 | 30 | 25 | 32
mIU/mL | -0.1 (1.0) | -2.4 (2.4) | 4.8 (4.7) | 6.9 (7.7)

3. Secondary Outcome: Change in FSH After 3 Months of Treatment
Time Frame: 3 months
Population: ITT population
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Placebo | Testim (Topical Testosterone) | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 26 | 30 | 25 | 32
mIU/mL | -0.2 (0.7) | -4.4 (2.9) | 5.1 (6.2) | 7.4 (6.5)

4. Secondary Outcome: Reproductive Safety
Description: Change from baseline in sperm concentration
Time Frame: 3 months
Population: Subjects with end of study assessments
Measure: Mean (Standard Deviation); unit: millions/mL
Arm/Group | Placebo | Testim (Topical Testosterone) | Androxal 12.5 mg | Androxal 25 mg
Number analyzed (Participants) | 13 | 13 | 12 | 19
millions/mL | -19.1 (93.4) | -29.5 (39.0) | 8.2 (233.1) | -2.8 (167.0)

ADVERSE EVENTS:
Arm/Group | Placebo | Testim (Topical Testosterone) | Androxal 12.5 mg | Androxal 25 mg
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/33 | 0/27 | 0/33
Other Adverse Events (participants affected / at risk) | 3/28 | 15/33 | 3/27 | 3/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Testim (Topical Testosterone) (N=33) | Androxal 12.5 mg (N=27) | Androxal 25 mg (N=33)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject was admitted to the hospital for high A1C level of 16.9. The PI assessed the event as moderate in intensity, and definitely not related to the study medication.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Testim (Topical Testosterone) (N=33) | Androxal 12.5 mg (N=27) | Androxal 25 mg (N=33)
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 1
Addominal Pain Upper (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0
Sperm concentration decreased (Investigations) | 0 | 8 | 0 | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication, Investigator shall submit to the Sponsor a copy of any proposed publication. Sponsor shall have sixty (60) days to review the proposed publication for possible disclosure of Sponsor's Confidential Information and, upon request of Sponsor, Investigator shall delete any of Sponsor's Confidential Information or withhold submission of such publication to allow Sponsor to protect its intellectual property rights.